CLINICAL TRIAL: NCT01179737
Title: A 24 Week, Randomized, Double Blind, Multicenter, Placebocontrolled Efficacy, Safety, Tolerability and PK Trial of Nilotinib (Tasigna®, AMN107) in Pulmonary Arterial Hypertension (PAH)
Brief Title: Efficacy, Safety, Tolerability and Pharmacokinetics (PK) of Nilotinib (AMN107) in Pulmonary Arterial Hypertension (PAH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to serious adverse event (SAE)
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAMN107X2201; 2010-019883-36 (EudraCT Number); NCT01531270 (obsolete NCT alias)
Record Dates: First submitted 2010-08-03; First posted 2010-08-11 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Nilotinib; 6MWD; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — nilotinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nilotinib (Experimental): Participants in cohort 1 were assigned to receive nilotinib 50 mg during 14 days, followed by 150 mg during 14 days, followed by 300 mg during 140 days. Participants in cohort 2 were assigned to receive nilotinib 300 mg during 168 days
  Interventions: Drug: Nilotinib
- Placebo (Placebo Comparator): Participants were assigned to receive placebo to nilotinib to match 50 mg and 150 mg capsules during 168 days.
  Interventions: Drug: Placebo to nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib capsules for oral administration at 50 mg, 150 mg twice a day and 300 mg (2 capsules of 150 mg) twice a day.
  Arms: Nilotinib
Drug: Placebo to nilotinib — Placebo to nilotinib capsules for oral administration to match 50 mg, 150 mg and 300 mg capsules twice a day
  Arms: Placebo

SUMMARY:
The purpose of this trial was to establish the safety, tolerability and PK of nilotinib in this population and to test the hypothesis that 6 months treatment with nilotinib will significantly reduce pulmonary artery resistance.

DETAILED DESCRIPTION:
The purpose of this trial was to establish the safety, tolerability and PK of nilotinib in this population and to test the hypothesis that 6 months

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO) Functional Class II or III
* 6MWD ≥ 150 m and ≤ 450 m at screening
* Current diagnosis of PAH according to Dana Point 2008 Meeting
* Inadequate clinical response on one or more class(es) of PAH drug
* Stabilization of pulmonary hypertension medications for ≥ 2 months on approved therapeutic dose of at least one PAH drug and still symptomatic with WHO functional Class II or III performance.

Exclusion Criteria:

* Women of child-bearing potential not practicing birth control
* In treatment with chronic nitric oxide therapy
* Pre-existing lung disease
* Use of drugs prolonging the QT interval or strong CYP3A4 inhibitors
* Long QT syndrome or QTc > 450 ms males; > 470 ms females.
* WHO Class IV
* Pulmonary capillary wedge pressure > 15 mm Hg
* Other diagnosis of PAH in WHO Diagnostic Group 1
* PAH associated with: venous hypertension (WHO Diagnostic Group II), hypoxia (WHO Diagnostic Group III), chronic pulmonary thromboembolic disease (WHO Diagnostic Group IV) or other miscellaneous causes (WHO Diagnostic Class V, which includes sarcoidosis, histiocytosis X, lymphangiomatosis, compression of pulmonary vessels)
* Thrombocytopenia < 50 x109/L (50 x 103/µL)
* Uncontrolled systemic arterial hypertension, systolic > 160 mm Hg or diastolic >90 mm Hg
* Any advanced, severe, or unstable disease of any type that may interfere with the primary and secondary endpoint evaluations.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (5):
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Nashville, Tennessee
- Novartis Investigative Site, Calgary, Alberta, Canada
- Germany (3):
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Marburg
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Zurich, Switzerland, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 participants were enrolled into the study (15 in cohort 1; 8 in cohort 2) 8 participants completed cohort 1 and 6 of these participants moved into cohort 1expansion. Of the 5 participants that completed Cohort 1 expansion; 3 participants went into an Extension. None of the participants completed treatment as trial was terminated
Pre-assignment Details: Participants were randomized 6:1 ratio to nilotinib and placebo
Groups:
- Cohort 1: Nilotinib: Participants were assigned to receive nilotinib 50 mg during 14 days, followed by 150 mg during 14 days, followed by 300 mg during 140 days.
- Cohort 1: Placebo: Participants were assigned to receive placebo to nilotinib to match 50 mg and 150 mg capsules during 168 days.
- Cohort 2: Nilotinib: Participants were assigned to receive nilotinib 300 mg during 168 days
- Cohort 2: Placebo: Participants were assigned to receive placebo to match 50mg and / or 150mg capsules during 168 days
Period: Cohort 1 & Cohort 2
Arm/Group | Cohort 1: Nilotinib | Cohort 1: Placebo | Cohort 2: Nilotinib | Cohort 2: Placebo
Started | 12 | 3 (One patient was missing the end of study evaluation) | 4 | 4
Completed | 7 | 1 | 0 | 0
Not Completed | 5 | 2 | 4 | 4
Not completed — Adverse Event | 3 | 1 | 1 | 0
Not completed — Withdrew consent | 2 | 0 | 0 | 0
Not completed — Administrative problems | 0 | 0 | 2 | 4
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Withdrew consent without EOS 1 visit | 0 | 1 | 0 | 0
Period: Cohort 1 & Cohort 2 Expansion
Arm/Group | Cohort 1: Nilotinib | Cohort 1: Placebo | Cohort 2: Nilotinib | Cohort 2: Placebo
Started | 5 (2 participants did not enroll in extension) | 1 | 0 | 0
Completed | 4 | 1 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Period: Extension
Arm/Group | Cohort 1: Nilotinib | Cohort 1: Placebo | Cohort 2: Nilotinib | Cohort 2: Placebo
Started | 3 (Two patients did not enrol in the extension) | 0 (One patient did not enrol in the extension) | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0
Not completed — The study was terminated | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: an end of study evaluation was only available for 14 of these patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Nilotinib | Cohort 1: Placebo | Cohort 2: Nilotinib | Cohort 2: Placebo | Total
Number analyzed (Participants) | 12 | 3 | 4 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52 (13.1) | 60 (6.1) | 31 (14.6) | 33 (10.2) | 32 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 4 | 3 | 20
  Male | 2 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Change in Six-Minute Walk Distance (6MWD) From Baseline
Description: During standardized walk course participants are connected to a portable pulse oximeter via a finger probe and instructed to walk at a comfortable speed for as far as they could manage in 6 minutes. Study was prematurely terminated and efficacy data were not analyzed or summarized
Time Frame: Baseline, 168 days
Groups:
- Change in Six-Minute Walk Distance (6MWD) From Baseline: During standardized walk course participants are connected to a portable pulse oximeter via a finger probe and instructed to walk at a comfortable speed for as far as they could manage in 6 minu
Arm/Group | Change in Six-Minute Walk Distance (6MWD) From Baseline
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Pulmonary Vascular Resistance (PVR)
Description: Change in pulmonary vascular resistance is measured via right heart catheter assessment according to local hospital procedures. It assesses several prognostic hemodynamic variables in pulmonary hypertension, including Pulmonary Vascular Resistance (PVR). Study was prematurely terminated and not powered for efficacy.
Time Frame: 168 days
Groups:
- Change in Pulmonary Vascular Resistance (PVR): Change in pulmonary vascular resistance is measured via right heart catheter assessment according to local hospital procedures. It assesses several prognostic hemodynamic variables in pulmonary hypertension, including Pulmonary Vascular Resistance (PVR).
  Additional information about the outcome measure, if needed for clarification. Outcome Measures are: Specific key measurement(s) or observation(s) used to measure the effect of experimental variables in a study, or for observational studies, to describe patterns of diseases or traits or associations with exposures, risk factors or treatment.
  Examples:
  Title: all cause mortality Time Frame: one year Safety Issue: No
  Title: Evidence of clinically definite ischemic stroke (focal neurological deficits persisting for more than 24 hours) confirmed by non-investigational CT or MRI Time Frame: within the first 30 days (plus or minus 3 days) after surgery Safety Issue: Yes
Arm/Group | Change in Pulmonary Vascular Resistance (PVR)
Number analyzed (Participants) | 0

3. Secondary Outcome: Total Number of Adverse Events and Serious Adverse Events
Description: Adverse events were summarized by the number of patients having any adverse event overall and presented in the safety section. Study was prematurely terminated.
Time Frame: 168 days
Groups:
- Total Number of Adverse Events and Serious Adverse Events: Adverse events were summarized by the number of patients having any adverse event overall and presented in the safety section.
Arm/Group | Total Number of Adverse Events and Serious Adverse Events
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the duration of treatment 140 days for cohort 1, 168 days for cohort 2 and up to 1092 days in the extension study
Description: 23 participants were enrolled into the study; 8 participants completed cohort 1 and 6 of these participants moved into cohort 1 expansion of which 5 participants completed Cohort 1 expansion. Of the 5 participants, 3 went into an Extension. None of the participants completed treatment as trial was terminated
Arm/Group | Cohort 1: Nilotinib | Cohort 1: Placebo | Cohort 2: Nilotinib | Cohort 2: Placebo
Serious Adverse Events (participants affected / at risk) | 7/12 | 1/3 | 2/4 | 1/4
Other Adverse Events (participants affected / at risk) | 12/12 | 1/3 | 3/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Nilotinib (N=12) | Cohort 1: Placebo (N=3) | Cohort 2: Nilotinib (N=4) | Cohort 2: Placebo (N=4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0
Torsade de pointes (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Device leakage (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 3 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0
Infusion site infection (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Nilotinib (N=12) | Cohort 1: Placebo (N=3) | Cohort 2: Nilotinib (N=4) | Cohort 2: Placebo (N=4)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Polychromasia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Red blood cell abnormality (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Dilatation ventricular (Cardiac disorders) | 2 | 0 | 0 | 0
Left atrial dilatation (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Right ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 3 | 0
Application site irritation (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0 | 0 | 0
Viral sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Biopsy bone (Investigations) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 0
Red blood cell burr cells present (Investigations) | 1 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 2 | 0 | 0 | 0
Right ventricular systolic pressure increased (Investigations) | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 1 | 3 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2
Decreased interest (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 1
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0
Inferior vena cava dilatation (Vascular disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety